CLINICAL TRIAL: NCT04096183
Title: Evaluation of Lung Volume Under Nasal High Flow With a Time of Flight Camera
Acronym: CamOpt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC19.0070_CamOpt
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: High Flow Nasal; Time of Flight Camera; Lung Volume; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ventilation of healthy volunteers (Other)
  Interventions: Other: Ventilation of healthy volunteers

INTERVENTIONS:
Other: Ventilation of healthy volunteers — Ventilation of healthy volunteers in different clinical situations

SUMMARY:
The effectiveness of Nasal High Flow therapy (NHF), in comparison with conventional oxygen therapy, is based on Positive Expiratory Pressure (PEP) and washout of dead space.

Many authors have shown that peak expiratory pressure, expiratory plateau pressure, mean upper airway pressure and lung volume were significantly increased. It depends mainly on gas flow and mouth closure.

First, "Groves"showed in 2007 that mouth opening could vary nasopharyngeal pressure from 2.7 to 7.4 cmH20 to 60 L / min, like Parke did in 2009, with a pressure of 1.2 at 2.7 cmH2O at 35 L / min.

Then, "Parke" showed in 2011 and 2015, a nasopharyngeal pressure changing from 2.7 to 11.9 cmH20 by varying the flow rate from 30 to 100 L / min. "Bräunlich" also showed concordant results in 2018, from 1.6 to 2.3 cmH2O, changing flow rates from 20 to 40 L / min. "Corley" in 2011 found a pressure from -0.3 to 2.7 by passing from ambient air to high flow. "Okuda and Mauri's" work in 2017 on oesophageal pressures also contributed to this.

In addition, it has been proved that the Tidal Volume (TV) is proportional to the flow delivered. These measurements were carried out by impedancemetry, the results of which were extrapolated to Vt. Thus "Okuda" evaluated it at 685mL in ambient air and 968mL at 50L / min. In 2016, "Fraser" highlighted a TV increasing from 400 to 500 mL by increasing the flow rate to 30 L / min. "Parke" in 2015 described an exponential End Expiratory Lung Impedence (EELI) proportional to the flow rate, as did "Riera" in 2013 with a ratio of 1.26 between ambient air and NHF at 40 L / min, and "Corley" in 2011 (ratio of 1.25).

Actualy, Time-of-Flight (ToF) cameras, such as Kinect v2®, are increasingly used in the medical field, particularly to characterize respiratory movement.

Various authors have shown a good correlation between the values of TV obtained by spirometry (reference method) and those obtained with ToF camera. A study led in 2018, by "S. Nazir" in the Department of "Réanimation Médicale" at the University Hospital of Brest, evaluated the average errors less than 46mL, with 76% of measurements having an error less than 50 mL, which corresponds to the clinical limit.

Now having a non-invasive, safe, simple, reproducible, inexpensive, and allowing evaluation in clinical situations method ; the use of a Time-of-Flight camera to evaluate the breathing and its various parameters, is indicated.

In this innovative study, never performed in different respiratory conditions in vigilant patients with NHF, the lung volume will be evaluated by a Time-of-Flight camera.

Different clinical situations, and the different parameters influencing it, will be observed and compared with the results of previous studies.

These situations will be simulations ranging from a physiological state to an acute respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and Major Volunteers

Exclusion Criteria:

* Nasopharyngeal obstruction, facial trauma, or other contraindication to the use of Nasal High Flow, pregnant woman, major incompetent, lack of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pulmonary volume change | 3 hours
  Changes on the pulmonary volume in different situations during 3 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be aviable for fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Le Moigne G, Nazir S, Pateau V, Courtois E, L'Her E. Noninvasive Tidal Volume Measurements, Using a Time-of-Flight Camera, Under High-Flow Nasal Cannula-A Physiological Evaluation, in Healthy Volunteers. Crit Care Med. 2022 Jan 1;50(1):e61-e70. doi: 10.1097/CCM.0000000000005183. PMID 34259664